CLINICAL TRIAL: NCT01995890
Title: Effect of Nepafenac Eye Drops on Intraocular Pressure - a Randomized Prospective Study
Brief Title: Effect of Nepafenac Eye Drops on Intraocular Pressure in Normal Eyes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr T V Patel Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TVPEI
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Intraocular Pressure
Keywords: nepafenac eye drops; intraocular pressure
MeSH Terms: interventions — nepafenac

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nepafenac (Experimental): Nepafenac 0.1% eye drops, 3 times a day
  Interventions: Drug: nepafenac
- control (No Intervention): No intervention in the control arm

INTERVENTIONS:
Drug: nepafenac
  Other Names: Nevanac
  Arms: nepafenac

SUMMARY:
The Nevanac product information insert says that it can cause increase in eye pressure in 5-10% of patients. There is very little published literature on the effect of topical Nepafenac eye drops on eye pressure in normal people. The purpose of our study is to report this effect with a working hypothesis that there is no increase in eye pressure following use of Nepafenac eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity better than 20/80 in both eyes
* Intraocular pressure ≤21 mmHg in both eyes
* Open angles on 4 mirror gonioscopy without indentation
* Normal optic disc on stereoscopic examination and photographs

Exclusion Criteria:

* Change in the systemic medication profile during the course of the study
* Allergy to nepafenac molecule
* Corneal thinning/corneal infections
* Any intraocular surgery in past 3 months
* Pregnancy or those planning to conceive
* Breast feeding patients
* Unwillingness to participate in the trial
* Concomitant use of any other ocular drug (except artificial tears)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 4 weeks
  Intraocular pressure elevation of more than 4 mmHg from baseline
Intraocular pressure | 8 weeks
  Intraocular pressure elevation of more than 4 mmHg from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paaraj R Dave, MD, Principal Investigator — TV Patel Eye Institute
Locations (1):
- Dr TV Patel Eye Insititute, Vadodara, Gujarat, India

REFERENCES:
- [Background] Gamache DA, Graff G, Brady MT, Spellman JM, Yanni JM. Nepafenac, a unique nonsteroidal prodrug with potential utility in the treatment of trauma-induced ocular inflammation: I. Assessment of anti-inflammatory efficacy. Inflammation. 2000 Aug;24(4):357-70. doi: 10.1023/a:1007049015148. PMID 10850857
- [Result] Chiba T, Kashiwagi K, Chiba N, Tsukahara S. Effect of non-steroidal anti-inflammatory ophthalmic solution on intraocular pressure reduction by latanoprost in patients with primary open angle glaucoma or ocular hypertension. Br J Ophthalmol. 2006 Mar;90(3):314-7. doi: 10.1136/bjo.2005.080895. PMID 16488953
- [Result] Warren KA, Fox JE. Topical nepafenac as an alternate treatment for cystoid macular edema in steroid responsive patients. Retina. 2008 Nov-Dec;28(10):1427-34. doi: 10.1097/IAE.0b013e31817e7ead. PMID 18664937